CLINICAL TRIAL: NCT03419195
Title: Cardiovascular Mechanisms of Exercise Intolerance in Diabetes and the Role of Sex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0356
Record Dates: First submitted 2018-01-18; First posted 2018-02-01 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes Mellitus; Healthy; Overweight; Cardiovascular Risk Factor
Keywords: Type 2 Diabetes; Overweight; Exercise Training; Exercise Impairment; Healthy Control; Veteran; Blood Flow
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 2 diabetes (Experimental): Men and women between the ages of 30-55 with well controlled type 2 diabetes (A1C <9%).
  Interventions: Other: Cardiovascular exercise training
- Healthy overweight controls (Experimental): Men and women between the ages of 30-55 with BMI 25-40 and limited immediate family history of type 2 diabetes.
  Interventions: Other: Cardiovascular exercise training

INTERVENTIONS:
Other: Cardiovascular exercise training — Following the completion of baseline testing, both subject groups will undergo supervised cardiovascular exercise training 3 times per week for 3 months (plus a 3 week ramp-up). Exercise training will take place on a treadmill, stationary bicycle, elliptical, rowing machine, or combination of machines. Each session will last 1 hour, which includes a 5 minute warm-up, 50 minutes of exercise, and a 5 minute cool down.
  Other Names: Exercise Training

SUMMARY:
This study will define the relationship of cardiac, vascular function and skeletal muscle blood flow (individually and together) to cardiovascular exercise capacity in in men and women with and without type 2 diabetes (T2DM). Identification of differences in the effects of exercise training on the integrated cardiovascular system and metabolism in men and women with and without T2DM will reveal specific adaptive responses to exercise.This study will evaluate & compare exercise function in a total of 60 subjects from the Denver area (30 people with T2DM and 30 overweight control subjects).

Specific Aim 1: To test the hypothesis that the integration of cardiac function, macrovascular function, and microvascular function is impaired in T2D and correlates with cardiovascular exercise capacity (CVEC) impairment.

Specific Aim 2: To test the hypothesis that exercise training will elicit adaptive responses in cardiac and vascular function, muscle perfusion and metabolism with differences by T2D status.

Differences between the exercise responses in people with T2DM and healthy people will help further identify the disease process of T2DM and direct future research of treatments and interventions.

DETAILED DESCRIPTION:
It is well established that functional exercise capacity and peak oxygen uptake (VO2) are reduced in patients with type 2 diabetes mellitus (T2DM) compared with healthy counterparts. The mechanisms underlying the exercise deficit in T2DM remain largely unknown, but previous work has suggested that reduced exercise blood flow and impaired submaximal VO2 may be contributing factors. Both of these findings are consistent with a peripheral impairment of skeletal muscle oxygen delivery, oxygen utilization, or both. Indeed, dysfunction of skeletal muscle metabolism plays a key role in the pathophysiology of T2DM, and considerable work has described abnormalities of oxidative function in the skeletal muscle of people with T2DM. Given this, it is likely that the causes of exercise intolerance in T2DM may relate to specific defects at the level of the skeletal muscle, particularly given that skeletal muscle blood flow and oxidative capacity are impaired in diabetes. However, to the knowledge of the investigators, no one has related these peripheral muscle abnormalities to the diminished exercise function in this patient group.

The overarching hypothesis for the proposed research is that impaired CVEC in T2DM is the result of preclinical cardiac, vascular dysfunction and skeletal muscle perfusion abnormalities. Exercise training will improve CVEC and will reveal specific reversible therapeutic aspects of this pathology. The investigators will first determine the impairments and then evaluate responses to an established cardiac rehabilitation exercise training program, established to improve fitness in people with and without diabetes. Given the greater CVEC abnormalities observed in women, sex differences will be evaluated for each aim.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with and without type 2 diabetes
* BMI 25-40
* Sedentary subjects not participating in a regular exercise program (<one bout of exercise/week)

Exclusion Criteria:

* Documented cardiovascular disease
* Uncontrolled hypertension: disease systolic blood pressure (SBP) > 150, diastolic blood pressure (DBP)> 110
* Obstructive pulmonary disease or asthma
* Peripheral neuropathy
* Physical impairment that would limit exercise ability
* Subjects taking beta blockers, calcium channel blockers, insulin, or Thiazolidinediones (TZD)
* Current or past smoking within the last 1 years
* Current tobacco use
* Anemia
* Control HbA1c > 5.7, T2DM HbA1c > 9
* Pregnant, nursing or hormonal therapy (other than contraceptives)
* Peri or post-menopausal women
* Type 1 diabetes
* Hepatic or renal disease.
* Peptic ulcer disease.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen consumption (VO2peak) | Through study completion, approximately 4 months
  Subjects' peak oxygen consumption will be tested on a stationary bike before and after 3 months of exercise
Change in insulin sensitivity | Through study completion, approximately 4 months
  The investigators will evaluate the changes in insulin sensitivity utilizing a euglycemic insulin clamp
Change in muscular mitochondrial function | Through study completion, approximately 4 months
  The investigators will examine mitochondrial function using magnetic resistance (MR) spectroscopy during single leg calf exercise

CONTACTS AND LOCATIONS:
Overall Officials: Judy Regensteiner, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park S, Englund EK, Fujiwara T, Enge D, Schafer M, Gerstner Saucedo J, Clark EW, Abushamat LA, Scalzo RL, Fonseca B, Hunter KS, Sammel MD, Regensteiner JG, Reusch JEB, Barker AJ. Comprehensive CMR evaluation including 4D flow-derived E/A vorticity ratio in overweight adults with and without type 2 diabetes mellitus. Cardiovasc Diabetol. 2025 Dec 8;25(1):7. doi: 10.1186/s12933-025-02999-9. PMID 41361416
- [Derived] Abushamat LA, Enge D, Fujiwara T, Schafer M, Clark EW, Englund EK, Scalzo RL, Johnston A, Rafferty D, Schauer IE, Whipple MO, Hunter K, Huebschmann AG, Nadeau KJ, Jarvis K, Barker AJ, Regensteiner JG, Reusch JEB. Obesity dominates early effects on cardiac structure and arterial stiffness in people with type 2 diabetes. J Hypertens. 2023 Nov 1;41(11):1775-1784. doi: 10.1097/HJH.0000000000003534. Epub 2023 Aug 17. PMID 37589719

DOCUMENTS (1):
  • Informed Consent Form (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT03419195/ICF_001.pdf